CLINICAL TRIAL: NCT02649439
Title: Prostvac in Patients With Biochemically Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160035; 16-C-0035
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer
Keywords: Vaccine; PSA; Surveillance; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A/PROSTVAC treatment (Experimental): PROSTVAC treatment for 6 months with an additional optional year of maintenance for eligible patients
  Interventions: Biological: PROSTVAC -V; Biological: PROSTVAC-F
- B/ Delayed PROSTVAC treatment (Experimental): Surveillance for 6 months followed by PROSTVAC treatment for 6 months with an additional year of maintenance for eligible patients
  Interventions: Biological: PROSTVAC -V; Biological: PROSTVAC-F

INTERVENTIONS:
Biological: PROSTVAC -V — Recombinant Vaccinia Virus Vector Vaccine of the Genus Orthopoxvirus
Biological: PROSTVAC-F — Recombinant Fowlpox Virus Vector Vaccine of the Genus Avipoxvirus

SUMMARY:
Background:

Some people who have been treated for prostate cancer still have high prostate-specific antigen (PSA) levels. This may indicate cancer. These people have non-metastatic castration sensitive prostate cancer (nmCSPC) or biochemical recurrent prostate cancer. Researchers think the immune system can be taught to fight and kill cancer cells. They think an immunotherapy vaccine called prostvac could help reduce PSA levels in people with this type of prostate cancer.

Objective:

To test if prostvac can decrease tumor growth rate as measured by PSA compared to getting surveillance alone.

Eligibility:

Men ages 18 or older who have nmCSPC or biochemical recurrent prostate cancer

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Bone scan

Computed tomography (CT) scan, or magnetic resonance imaging (MRI) and positron emission tomography (PET) scan: They lie in a machine that takes pictures of the body.

Electrocardiogram: Soft electrodes are stuck to the skin to record heart signals.

Participants will be part of 1 of 2 arms: Arm A will get prostvac for 6 months. Arm B will have surveillance for 6 months followed by prostvac for 6 months.

During the prostvac period, participants will get prostvac as a shot under the skin on weeks 1, 3, and 5, and then monthly for a total of 5 months.

Participants will have follow-up visits at least every month until they recover from prostvac side effects or their cancer worsens. Visits may include repeats of screening tests.

Participants will be followed for up to 15 years. They will have a physical exam every year for the first 5 years. They will have phone calls once a year.

DETAILED DESCRIPTION:
BACKGROUND

* Androgen deprivation therapy (ADT) and surveillance are treatment options for prostate cancer patients with biochemical progression after localized therapy (biochemically recurrent prostate cancer). The primary goal in these patients is to prevent morbidity from their cancer and to do so with limited toxicity.
* Prostvac (Prostvac; developed by the National Cancer Institute [NCI] and licensed to BN Immunotherapeutics, Mountain View, CA) is a novel candidate prostate cancer immunotherapy for the treatment of prostate cancer. It is a viral vector based therapeutic cancer vaccine that is administered via subcutaneous injections. In a randomized controlled Phase 2 trial, Prostvac therapy was associated with a prolongation of survival in men with metastatic castrate-resistant prostate cancer. A phase III trial recently completed accrual of patients in this same population.
* There is also rationale to use therapeutic cancer vaccines such as Prostvac in earlier stage prostate cancer patients to maximize the potential therapeutic effect of immune stimulating therapy.
* Analysis of previous trials using therapeutic cancer vaccines alone suggests that such therapies may alter tumor growth rate.

OBJECTIVE

Primary Objective:

-Determine if the therapeutic cancer vaccine prostvac can decrease tumor growth rate as measured by prostate-specific antigen (PSA) rise after 6 months compared to a group getting surveillance alone.

KEY ELIGIBILITY CRITERIA

* Histologically confirmed adenocarcinoma of the prostate
* Patients with negative computed tomography (CT) Scan and Tc-99m Bone Scan
* Patients with a PSA over 0.8 ng/ml for patients following radical prostatectomy or for patients following definitive radiation therapy: a rise in PSA of greater than or equal to 2 ng/mL above the nadir
* Patients with a PSA doubling time of 5-15 months
* No history of active autoimmune disease or history of organ compromising autoimmune disease
* Eastern Cooperative Oncology Group (ECOG) 0 -1

DESIGN

* Randomized study
* Accrual goal is 36 evaluable patients per arm; randomized 1:1 to:

  * Arm A: Prostvac for 6 months with an additional optional year of maintenance for eligible patients OR
  * Arm B: Surveillance for 6 months, then Prostvac for 6 months with an additional year of maintenance for eligible patients

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histopathological documentation of prostate cancer confirmed in either the Laboratory of Pathology at the National Institutes of Health (NIH) Clinical Center, Walter Reed National Military Medical Center, Memorial Sloan Kettering Cancer Center (MSKCC), Dana-Farber Cancer Institute (DFCI) or Beth Israel Deaconess Medical Center (BIDMC) prior to enrollment. If no pathologic specimen is available, patients may enroll with a pathologists report showing a histologic diagnosis of prostate cancer and a clinical course consistent with the disease.
* Biochemical progression after definitive radiation or surgery defined as follows:

  * For patients following definitive therapy: a rise in prostate-specific antigen (PSA) of greater than or equal to 2ng/mL above the nadir (per Radiation Therapy Oncology Group (RTOG)-American Society for Therapeutic Radiology and Oncology (ASTRO) consensus criteria).
  * For patients following radical prostatectomy: rising PSA after surgical procedure. (Patients must have a PSA greater than or equal to 0.8 ng/ml)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 1 (Karnofsky greater than or equal to 80%).
* Patients must have a PSA doubling time of 5-15 months.
* Patients must have a rising PSA as confirmed by 3 values done at least 1 week apart and over no less than 1 month.
* Recovery from acute toxicity related to prior therapy, including surgery and radiation, or no toxicity greater than or equal to grade 2.
* Negative computed tomography (CT) scan/magnetic resonance imaging (MRI) and bone scan for metastatic prostate cancer.
* Hematological eligibility parameters (within 16 days before starting therapy)

  * Granulocyte count greater than or equal to 1000/mm^3
  * Platelet count greater than or equal to 100 000/mm^3
  * Hemoglobin (Hgb) greater than or equal to 10g/dL
* Biochemical eligibility parameters (within 16 days before starting therapy):

  --Hepatic function: bilirubin less than or equal to 1.5mg/dL (OR in patients with Gilbert's syndrome normal.
* No other active malignancies within the past 36 months (with the exception of nonmelanoma skin cancers or carcinoma in situ of the bladder) or life-threatening illnesses, in the opinion of the investigator
* Willing to travel to the National Institutes of Health (NIH), MSKCC, DFCI, BIDMC for follow-up visits.
* 18 years of age or older.
* Able to understand and sign informed consent.
* Baseline testosterone greater than or equal to 100 ng/dl
* PSA less than or equal to 30 ng/mL.
* The effects PROSTVAC on the developing human fetus are unknown. For this reason, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study therapy and at least one month post therapy. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Immunocompromised status due to:

  * Human immunodeficiency virus (HIV) positivity.
  * Active autoimmune diseases such as Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome or active Grave's disease. Patients with a history of autoimmunity that has not required systemic immunosuppressive therapy or does not threaten vital organ function including central nervous system (CNS), heart, lungs, kidneys, skin, and gastrointestinal (GI) tract will be allowed.
  * Other immunodeficiency diseases
  * Splenectomy
* Chronic administration (defined as daily or every other day for continued use > 14 days) of corticosteroids deemed systemic by investigator within 28 days before the first planned dose of PROSTVAC. Use of inhaled steroids, nasal sprays, intra-articular injections and topical creams for small body areas is allowed.
* Serious intercurrent medical illness that, in the judgment of the investigator, would interfere with patient s ability to carry out the treatment program.
* Other medications used for urinary symptoms including 5-alpha reductase inhibitors (finasteride and dutasteride) and alternative medications known to alter PSA (eg phytoestrogens and saw palmetto)
* History of prior chemotherapy
* History of prior immunotherapy within the last 3 years
* Major surgery within 4 weeks prior to enrollment (Day 1 visit).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to poxviral vaccines (e.g., vaccinia vaccine)
* Known allergy to eggs, egg products, aminoglycoside antibiotics (for example, gentamicin or tobramycin).
* History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis
* Previous serious adverse reactions to smallpox vaccination
* Unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the Day 1 vaccination: Day 1 vaccination: (a) children less than or equal to 3 years of age, (b) pregnant or nursing women, (c) individuals with current or extensive eczema or other eczemoid skin disorders, or (d) immunocompromised individuals, such as those with HIV.
* Receipt of an investigational agent within 28 days (or 56 days for an antibody-based therapy) before the first planned dose of study drugs.
* Patients who test positive for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Uncontrolled hypertension (systolic blood pressure (SBP)>170/ DBP>105)
* Recruitment Strategies

This study will be listed on available websites (www.clinicaltrials.gov,

https://ccr.cancer.gov/clinical-trials-search-start) and participants will be recruited from the current patient population at NIH.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0035.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 97 participants were enrolled and 17/97 were screen failures who were enrolled and not treated. They are not included in the table because "potential participants who are screened for the purpose of determining eligibility, but do not participate, are not considered enrolled unless otherwise specified by the protocol", and that is not otherwise specified in the protocol.
Period: Overall Study
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment
Started | 40 | 40
Completed | 13 | 12
Not Completed | 27 | 28
Not completed — Switched to alternative treatment | 6 | 4
Not completed — Patient decision | 1 | 0
Not completed — Patient going out of country | 1 | 0
Not completed — To start finasteride | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Disease progression on study | 12 | 13
Not completed — Refused further treatment | 1 | 0
Not completed — Refused further follow up | 2 | 7
Not completed — Completed treatment phase but refused the protocol specified follow up | 1 | 0
Not completed — No treatment, per protocol | 1 | 0
Not completed — PSA DT makes ineligible | 0 | 1
Not completed — Rising PSA No Mets | 0 | 1
Not completed — Rising PSA | 0 | 1
Not completed — Signed follow up protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 18 | 30
  >=65 years | 28 | 22 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.06 (6.48) | 67.02 (6.56) | 67.04 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 33 | 32 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Median Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/ml] — Normal PSA is zero.
  ng/ml | 2.98 [0.83 to 28.15] | 2.82 [0.95 to 19.39] | 2.9 [0.89 to 23.77]

OUTCOME MEASURES:

1. Primary Outcome: Tumor Growth Rate as Measured by Prostate-specific Antigen (PSA) Rise After 6 Months When PROSTVAC is Initiated Compared to a Group on Surveillance for 6 Months
Description: Tumor growth rate was measured using the equation PSA (log growth rate) +/- SE (standard error).
Time Frame: 6 months
Measure: Number; unit: Unitless
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment
Number analyzed (Participants) | 40 | 40
Unitless | -2.528 | -2.449
Statistical Analysis 1: Comparison: A/PROSTVAC Treatment vs B/ Delayed PROSTVAC Treatment; Test type: Superiority; p = 0.4852, Wilcoxon signed rank test

2. Secondary Outcome: Effects of Vaccine on Prostate-specific Antigen (PSA) Growth Rate When PROSTVAC is Initiated After 6 Months on Surveillance
Description: Tumor growth rate was measured using the equation PSA (log growth rate) +/- SE (standard error).
Time Frame: After the participants in the Arm/Group "B/ Delayed PROSTVAC Treatment" received treatment for 6 months after their 6 month surveillance (e.g., 12 months total).
Population: 33/40 were evaluable in the first group.
Measure: Number; unit: Unitless
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment
Number analyzed (Participants) | 33 | 40
Unitless | -2.513 | -2.449
Statistical Analysis 1: Comparison: A/PROSTVAC Treatment vs B/ Delayed PROSTVAC Treatment; Test type: Superiority; p = 0.3269, Wilcoxon signed rank test

3. Secondary Outcome: Number of Participants With Prostate-specific Antigen (PSA) Specific T-Cells at Baseline and 6 Months
Description: Normal PSA is 0 nanograms per milliliter (ng/mL). Above 0 ng/mL is considered an increase in tumor growth.
Time Frame: Baseline and 6 months
Population: 35/40 and 32/40 participants are reported because these are the numbers of participants with sufficient samples for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment
Number analyzed (Participants) | 35 | 32
Participants
  Baseline | 22 | 20
  6 Months | 14 | 11

4. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 55 months and 13 days for Arm/Group A, and 57 months and 22 days for Arm/Group B.
Measure: Count of Participants; unit: Participants
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment
Number analyzed (Participants) | 40 | 40
Participants | 40 | 39

5. Other Pre Specified Outcome: Median Late Change in Peripheral Blood Mononuclear Cells (PBMCs) in Refined Subsets Monocyte Nonclassical, Monocyte Nonclassical Programmed Death Ligand 1 (PD-L1+), and Monocyte PD-1+ After PROSTVAC
Description: Blood samples collected were analyzed by multicolor flow cytometry in PBMCs for refined subsets of Monocytes. Changes in levels of PBMC subsets was a descriptive result with median percent change and interquartile range reported. P values were calculated using the Mann Whitney Test.
Time Frame: Day 29 (Post vaccination) vs Pre (Baseline)
Population: 7/40 and 29/40 participants were evaluable in the first and second group, respectively, based on availability of peripheral blood mononuclear cells (PBMCs) before and after vaccination.
Measure: Median (Inter-Quartile Range); unit: Percent change
Groups:
- A/PROSTVAC Treatment Responders; B/ Delayed PROSTVAC Treatment Non-Responders: PROSTVAC treatment for 6 months with an additional optional year of maintenance for eligible patients
  PROSTVAC -V: Recombinant Vaccinia Virus Vector Vaccine of the Genus Orthopoxvirus
  PROSTVAC-F: Recombinant Fowlpox Virus Vector Vaccine of the Genus Avipoxvirus
Arm/Group | A/PROSTVAC Treatment Responders | B/ Delayed PROSTVAC Treatment Non-Responders
Number analyzed (Participants) | 7 | 29
Percent change
  Monocyte Nonclassical Refined Subset | -29.8 [-70.8 to 10.0] | 9.3 [-26.6 to 41.4]
  Monocyte Nonclassical PD-L1+ Refined Subset | -57.5 [-73.7 to -2.8] | 17.3 [-15.1 to 56.5]
  Monocyte PD-1+ Refined Subset | -55.7 [-73.1 to -8.2] | -17.2 [-38.8 to 15.9]
Statistical Analysis 1: Comparison: A/PROSTVAC Treatment Responders vs B/ Delayed PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.0255, Mann Whitney Test — The reported p-value is representative of the PBMCs in monocyte nonclassical between responders and non-responders
Statistical Analysis 2: Comparison: A/PROSTVAC Treatment Responders vs B/ Delayed PROSTVAC Treatment Non-Responders; Test type: Other; p = 0.0021, Mann Whitney Test — The reported p-value is representative of the PBMCs in monocyte nonclassical PD-L1+ between responders and non-responders
Statistical Analysis 3: Comparison: A/PROSTVAC Treatment Responders vs B/ Delayed PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.0486, Mann Whitney Test — The reported p-value is representative of the PBMCs in monocyte PD-1+ between responders and non-responders

6. Other Pre Specified Outcome: Median Late Change in Peripheral Blood Mononuclear Cells (PBMCs) in Cluster of Differentiation 4 (CD4), Cluster of Differentiation 8 (CD8), Regulatory T-cells (Treg), Natural Killer (NK), and Myeloid-derived Suppressor Cells (MDSC) After PROSTVAC
Description: Blood samples collected were analyzed by multicolor flow cytometry in PBMCs for cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), Natural Killer (NK), myeloid-derived suppressor cell (MDSC) and Tregs. P values were calculated using the Mann Whitney Test.
Time Frame: Day 29 (Post vaccination) vs Pre (Baseline)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Percent change
Groups:
- A/PROSTVAC Treatment Non-Responders: PROSTVAC treatment for 6 months with an additional optional year of maintenance for eligible patients
  PROSTVAC -V: Recombinant Vaccinia Virus Vector Vaccine of the Genus Orthopoxvirus
  PROSTVAC-F: Recombinant Fowlpox Virus Vector Vaccine of the Genus Avipoxvirus
Arm/Group | A/PROSTVAC Treatment Responders | A/PROSTVAC Treatment Non-Responders
Number analyzed (Participants) | 7 | 29
Percent change
  Classic Subset CD4 | -7.1 [-51.7 to 13.0] | -3.3 [-13.4 to 11.2]
  Classic Subset CD8 | 1.2 [-16.9 to 51.8] | 2.8 [-12.0 to 15.2]
  Classic Subset Treg | 44.7 [-24.8 to 54.2] | 0.7 [-23.7 to 46.2]
  Classic Subset NK | 26.2 [-8.7 to 72.0] | 24.1 [-1.7 to 51.7]
  Classic Subset MDSC | 39.5 [-67.6 to 680.1] | 20.9 [-12.6 to 118.5]
Statistical Analysis 1: Comparison: A/PROSTVAC Treatment Responders vs A/PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.7317, Mann Whitney Test — The reported p-value is representative of the PBMCs in CD4 between responders and non-responders
Statistical Analysis 2: Comparison: A/PROSTVAC Treatment Responders vs A/PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.7545, Mann Whitney Test — The reported p-value is representative of the PBMCs in CD8 between responders and non-responders
Statistical Analysis 3: Comparison: A/PROSTVAC Treatment Responders vs A/PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.5310, Mann Whitney Test — The reported p-value is representative of the PBMCs in Treg between responders and non-responders
Statistical Analysis 4: Comparison: A/PROSTVAC Treatment Responders vs A/PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.8451, Mann Whitney Test — The reported p-value is representative of the PBMCs in NK between responders and non-responders
Statistical Analysis 5: Comparison: A/PROSTVAC Treatment Responders vs A/PROSTVAC Treatment Non-Responders; Test type: Superiority; p = 0.9377, Mann Whitney Test — The reported p-value is representative of the PBMCs in MDSC between responders and non-responders

7. Other Pre Specified Outcome: Peripheral Blood Mononuclear Cells (PBMCs) in Cluster of Differentiation 4 (CD4), Cluster of Differentiation 8 (CD8), Regulatory T-cells (Treg), Natural Killer (NK), and Myeloid-derived Suppressor Cells (MDSC), and naïve CD4 and CD8 T Cells After PROSTVAC
Description: Blood samples collected were analyzed by multicolor flow cytometry in PBMCs for cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), Natural Killer (NK), myeloid-derived suppressor cell (MDSC), Tregs, and naïve CD4 and naïve CD8 T cells. P values were calculated using the Wilcoxon signed rank test.
Time Frame: Baseline (Day 1) and one month (Day 29) after vaccine or surveillance (in the Delayed PROSTVAC group)
Population: 36 and 12participants were evaluable in the first and second group, respectively, based on availability of peripheral blood mononuclear cells (PBMCs) before and after vaccination or surveillance (in the Delayed PROSTVAC group).
Measure: Median (Inter-Quartile Range); unit: Percentage of PBMC
Groups:
- A/PROSTVAC Treatment Day 1; A/PROSTVAC Treatment Day 29: PROSTVAC treatment for 6 months with an additional optional year of maintenance for eligible patients
  PROSTVAC -V: Recombinant Vaccinia Virus Vector Vaccine of the Genus Orthopoxvirus
  PROSTVAC-F: Recombinant Fowlpox Virus Vector Vaccine of the Genus Avipoxvirus
- B/ Delayed PROSTVAC Treatment Day 1; B/ Delayed PROSTVAC Treatment Day 29: Surveillance for 6 months followed by PROSTVAC treatment for 6 months with an additional year of maintenance for eligible patients
  PROSTVAC -V: Recombinant Vaccinia Virus Vector Vaccine of the Genus Orthopoxvirus
  PROSTVAC-F: Recombinant Fowlpox Virus Vector Vaccine of the Genus Avipoxvirus
Arm/Group | A/PROSTVAC Treatment Day 1 | A/PROSTVAC Treatment Day 29 | B/ Delayed PROSTVAC Treatment Day 1 | B/ Delayed PROSTVAC Treatment Day 29
Number analyzed (Participants) | 36 | 36 | 12 | 12
Percentage of PBMC
  CD4 | 29.83 [25.04 to 39.98] | 29.16 [23.69 to 35.07] | 32.44 [27.37 to 34.72] | 29.07 [26.86 to 36.25]
  CD8 | 8.87 [6.97 to 13.34] | 9.98 [6.96 to 15.28] | 12.71 [8.78 to 18.54] | 13.00 [8.65 to 18.55]
  Treg | 0.58 [0.39 to 0.82] | 0.59 [0.49 to 0.96] | 1.03 [0.76 to 1.25] | 0.99 [0.67 to 1.25]
  NK | 8.04 [5.64 to 9.08] | 9.28 [5.79 to 14.39] | 10.35 [5.82 to 16.03] | 10.17 [6.18 to 15.93]
  MDSC | 4.60 [1.83 to 8.75] | 6.02 [3.19 to 9.00] | 5.74 [2.42 to 7.28] | 5.52 [3.06 to 7.32]
  Naive CD4 | 7.23 [3.11 to 10.13] | 6.93 [2.77 to 12.07] | 7.44 [2.93 to 11.27] | 7.12 [3.58 to 9.09]
  Naïve CD8 | 1.51 [0.81 to 2.72] | 1.26 [0.83 to 2.71] | 1.54 [0.60 to 3.84] | 1.39 [0.77 to 3.39]
Statistical Analysis 1: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.2012, Wilcoxon signed rank test — The reported p-value is representative of the % of CD4 in PBMCs at Day 1 and Day 29
Statistical Analysis 2: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.4891, Wilcoxon signed rank test — The reported p-value is representative of the % of CD8 in PBMCs at Day 1 and Day 29
Statistical Analysis 3: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.4609, Wilcoxon signed rank test — The reported p-value is representative of the % of Tregs in PBMCs at Day 1 and Day 29
Statistical Analysis 4: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.0012, Wilcoxon signed rank test — The reported p-value is representative of the % of NK in PBMCs at Day 1 and Day 29
Statistical Analysis 5: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.0825, Wilcoxon signed rank test — The reported p-value is representative of the % of MDSC in PBMCs at Day 1 and Day 29
Statistical Analysis 6: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.5988, Wilcoxon signed rank test — The reported p-value is representative of the % of naïve CD4 in PBMCs at Day 1 and Day 29
Statistical Analysis 7: Comparison: A/PROSTVAC Treatment Day 1 vs A/PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.5920, Wilcoxon signed rank test; The reported p-value is representative of the % of naïve CD8 in PBMCs at Day 1 and Day 29
Statistical Analysis 8: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.6221, Wilcoxon signed rank test — The reported p-value is representative of the % of CD4 in PBMCs at Day 1 and Day 29
Statistical Analysis 9: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.7334, Wilcoxon signed rank test — The reported p-value is representative of the % of CD8 in PBMCs at Day 1 and Day 29
Statistical Analysis 10: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Other; p = 0.7910, Wilcoxon signed rank test — The reported p-value is representative of the % of Tregs in PBMCs at Day 1 and Day 29
Statistical Analysis 11: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.5186, Wilcoxon signed rank test — The reported p-value is representative of the % of NK in PBMCs at Day 1 and Day 29
Statistical Analysis 12: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Superiority — The reported p-value is representative of the % of MDSC in PBMCs at Day 1 and Day 29; p = 0.5186, Wilcoxon signed rank test
Statistical Analysis 13: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.9097, Wilcoxon signed rank test — The reported p-value is representative of the % of naïve CD4 in PBMCs at Day 1 and Day 29
Statistical Analysis 14: Comparison: B/ Delayed PROSTVAC Treatment Day 1 vs B/ Delayed PROSTVAC Treatment Day 29; Test type: Superiority; p = 0.7334, Wilcoxon signed rank test — The reported p-value is representative of the % of naïve CD8 in PBMCs at Day 1 and Day 29

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 55 months and 13 days for Arm/Group A, and 57 months and 22 days for Arm/Group B.
Arm/Group | A/PROSTVAC Treatment | B/ Delayed PROSTVAC Treatment
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 3/40 | 6/40
Other Adverse Events (participants affected / at risk) | 40/40 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/PROSTVAC Treatment (N=40) | B/ Delayed PROSTVAC Treatment (N=40)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, Viral Myocarditis (Infections and infestations) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/PROSTVAC Treatment (N=40) | B/ Delayed PROSTVAC Treatment (N=40)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Aspartate aminotransferase increased (Psychiatric disorders) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Creatinine increased (Investigations) | 2 (4) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fatigue (General disorders) | 11 (13) | 16 (19)
Fever (General disorders) | 3 (3) | 2 (2)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 2 (2) | 1 (1)
Flu like symptoms (General disorders) | 6 (8) | 6 (10)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Infections and infestations) | 3 (5) | 5 (5)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3) | 4 (5)
Hemorrhagic episode of left eye (Eye disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (9) | 2 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 11 (12) | 9 (18)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (12) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 29 (119) | 33 (85)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 2 (5)
Malaise (General disorders) | 4 (4) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3)
Pain (General disorders) | 9 (10) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in left heel (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (6)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 2 (4) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Weight gain (Investigations) | 1 (1) | 1 (2)
Weight loss (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT02649439/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02649439/ICF_001.pdf